CLINICAL TRIAL: NCT04799925
Title: Effect of Treatment of Hyperuricemia on Progression of Diabetic Nephropathy in Patients With Type II Diabetes Mellitus and Stage III Chronic Kidney Disease.
Brief Title: Hyperuricemia and Diabetic Nephropathy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, mohammad ragab eldremi, Principal Investigator, Assiut University
Other Study IDs: Diabetic Nephropathy Uric Acid
Record Dates: First submitted 2021-03-05; First posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Hyperuricemia; Diabetic Nephropathies
MeSH Terms: conditions — Hyperuricemia; Diabetic Nephropathies | interventions — Febuxostat

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention group: Hyperuricemic group will be treated with uric acid lowering drug (febuxostat 80 mg once daily for 6 months).
  Interventions: Drug: Febuxostat
- Placebo group: Hyperuricemic group will take placebo pills.

INTERVENTIONS:
Drug: Febuxostat — uric acid lowering agent. dose: 80 mg once daily. duration: for 6 months
  Groups: Intervention group

SUMMARY:
The purpose of the study is to detect the effect of treatment of hyperuricemia on eGFR (Estimated Glomerular Filtration Rate) as an objective criterion for assessment of progression of diabetic nephropathy in patients with Type 2 Diabetes Mellitus.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will undergo a 1-week screening period to determine eligibility for study entry.

At week 0, patients who meet the eligibility requirements will be randomized in a double-blind manner (participant and investigator) in a 1:1 ratio to Febuxostat (80 mg, once daily) or Placebo (once daily) in patients with Type 2 Diabetes Mellitus and Stage 3 Chronic Kidney Disease (Estimated Glomerular Filtration Rate 31:59).

ELIGIBILITY:
Inclusion Criteria:

* Patient population will include both males and females above the age of 18 years with T2DM and Diabetic Nephropathy stage 3 CKD (eGFR: 31-59).

Exclusion Criteria:

* Patients with history of hypothyroidism, alcoholism, urinary tract infections, glomerulonephritis, myeloproliferative disorders and gout "as gout is a common inflammatory arthropathy characterized by painful and swollen joints resulting from precipitating uric acid crystals but hyperuricemia is commonly asymptomatic" or on drugs capable of inducing Hyperuricemia will be excluded from the study.
* Any patient will develop acute kidney injury episode at any time of the study will be excluded from the study.
* Patients with uncontrolled hypertension will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient population will include both males and females above the age of 18 years with T2DM and Diabetic Nephropathy stage 3 CKD (eGFR: 31-59).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-04-15 (Estimated); Primary Completion 2022-04-15 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Effect of treatment of hyperuricemia on estimated Glomerular Filtration Rate by the CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) equation. | 6 months from September 2021 to march 2022.
  Number of Participants with type 2 Diabetes Mellitus and stage 3 Chronic Kidney Disease (eGFR: 31:59) will be treated with uric acid lowering drug (febuxostat, 80 mg, once daily) for 6 months to detect the effect of treatment of hyperuricemia on estimated Glomerular Filtration Rate by the CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) equation.

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-02-20): https://cdn.clinicaltrials.gov/large-docs/25/NCT04799925/Prot_SAP_ICF_000.pdf